CLINICAL TRIAL: NCT00207337
Title: A Prospective Feasibility Study to Evaluate the Safety and Performance of the Exhale(R) Drug-Eluting Stent System in Patients With Emphysema
Brief Title: Exhale (R) Stent for Emphysema
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Broncus Technologies (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0304-28
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2008-01-23 (Estimated); Status verified 2008-01

CONDITIONS: Emphysema
Keywords: COPD (Chronic Obstructive Pulmonary Disease); Emphysema; Minimally invasive
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Device: Exhale Drug-Eluting Stent

SUMMARY:
Current treatment for emphysema is limited to measures that include inhaled oxygen, bronchodilators, anti-inflammatory drugs and pulmonary rehabilitation. Highly invasive procedures such as lung volume reduction surgery or lung transplantation are also performed. Treatment using the Exhale Drug-Eluting Stent (DES) is a minimally invasive bronchoscopic treatment that has the potential to reduce shortness of breath in emphysema patients. This study tests the safety and effects of Exhale DES in the treatment of patients with emphysema.

DETAILED DESCRIPTION:
Emphysema affects an estimated 60 million people worldwide and is a major cause of morbidity and mortality. In its most basic terms, emphysema causes the destruction of lung parenchyma resulting in collateral ventilation from one part of the lung to another through the disrupted alveolar walls, to the point that gas transport from one part of the lung to another may exceed gas flow through the small airways. In other words, the gas can move freely about within the lung, but it cannot get out, which causes over inflation, or hyperinflation of the diseased lung. When the disease is far advanced, patients are afflicted with disabling dyspnea that progressively restricts their activities and eventually causes great suffering. The crippling effects of end-stage emphysema, including severe dyspnea and marked limitation of activities, relate in large measure to the dynamic hyperinflation of the lungs associated with the loss of elasticity, gas trapping and collapse of small airways. The progressive enlargement of the thorax and flattening of the diaphragm render inspiratory muscles inefficient, increase the work of breathing and contribute to a feeling of breathlessness. The major medical therapeutic modalities include bronchodilator and anti-inflammatory drugs directed at decreasing airway resistance and antibiotics to combat infection. Pulmonary rehabilitation techniques and exercise training have proven of palliative benefit. In general, the results of medical treatment for advanced airway obstruction frequently result in a persistently anguished patient and frustrated physician. A system that could efficiently decompress emphysematous lungs with each breath would result in significant clinical benefit, including lessened dyspnea, decreased work of breathing, and increased exercise tolerance.

In addition to medical therapies, there are two surgical therapies available to emphysema sufferers: Lung transplantation and Lung Volume Reduction Surgery (LVRS). In the National Emphysema Treatment Trial (NETT), LVRS was shown to be effective in a sub-set of emphysema patients, but it had the drawback of increased short-term mortality as compared to the medical control arm. This was likely due to the invasiveness of LVRS.

Lung transplantation is a widely accepted surgical treatment for emphysema; however it is an unrealistic option for most patients. The selection criteria are very stringent for acceptance to receive a donor lung(s). Lung transplantation carries a high long-term morbidity and mortality and is severely limited by the shortage of available donor lungs.

We seek to take advantage of collateral ventilation seen in advanced emphysema by creating passageways from the lung parenchyma to large airways, through which air can escape the lungs during exhalation. The Exhale therapeutic intervention should be applicable to the majority of emphysema patients who suffer from hyperinflation of their lungs. It would be desirable to have a therapeutic option that is both less invasive and more readily available to emphysema sufferers. We have been working on such a therapy and have begun to investigate it in the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. High resolution computed tomography (CT) scan evidence of bilateral emphysema
2. Residual volume (RV) ≥ 220% predicted.
3. Total lung capacity (TLC) ≥ 133% of predicted value.
4. Forced expiratory volume (FEV1) < 40% of predicted or FEV1 < 1 liter.
5. Marked dyspnea, scoring ≥ 2 on the modified Medical Research Council scale of 0-4.
6. Patient has undergone pulmonary rehabilitation of 16 - 20 sessions.

Exclusion Criteria:

1. FEV1 > 20%
2. Diffusing capacity for carbon monoxide (DLco) < 15% of predicted.
3. Respiratory infection requiring > 3 hospitalizations in past year
4. Inability to walk > 140 meters in 6 minutes
5. Giant bulla > 1/3 of one lung's volume
6. Previous lung volume reduction surgery (LVRS) or lobectomy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-07; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Procedural and technical success - operatively
Decrease in residual volume > 300mL from baseline
Safety

SECONDARY OUTCOMES:
Dyspnea scoring
Pulmonary function measures
Exercise tolerance
Quality of life measures

CONTACTS AND LOCATIONS:
Overall Officials: Gregory I. Snell, MD, Principal Investigator — The Alfred
Locations (6):
- Australia (3):
  - The Prince Charles Hospital, Rode Road, Chermside, Queensland
  - The Alfred Hospital, Prahran, Victoria
  - Concord Repatriation General Hospital, Burwood
- Irmandade Santa Casa de Misericordia, Porto Alegre, Brazil
- Germany (2):
  - Universitätsklinik des Saarlandes, Homburg, Saarland
  - Medizinische Hochschule Hannover, Hanover

REFERENCES:
- See also: Broncus Technologies, Inc corporate web page — http://www.broncus.com
- See also: American Lung Association — http://www.lungusa.org